CLINICAL TRIAL: NCT05375643
Title: SURGE: Supporting UnderRepresented Minorities in Genomics-based Cancer Trial Enrollment (Intervention)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nadine McCleary, MD, MPH (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Nadine McCleary, MD, MPH, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-709
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Cancer; Hematologic Cancer; Thoracic Cancer
Keywords: Gastrointestinal Cancer; Hematologic Cancer; Thoracic Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm B (informational video) (Experimental): Participants will complete screening questionnaire via text or by phone to establish baseline awareness and interest in clinical trials and then randomized to the SURGE intervention where they will receive:
  * Informational Video
  Interventions: Behavioral: SURGE
- Arm A (standard of care) (No Intervention): Participants will complete screening questionnaire via text or by phone to establish baseline awareness and interest in clinical trials and then randomized to Standard of Care (SOC) and receive:
  * Standard of Care
- Arm C (informational video and patient navigation) (Experimental): Participants will complete screening questionnaire via text or by phone to establish baseline awareness and interest in clinical trials and then randomized to the SURGE intervention where they will receive:
  * Informational Video and Patient Navigation
  Interventions: Behavioral: SURGE

INTERVENTIONS:
Behavioral: SURGE — Video with or without person to person guidance to support decision making around genetic testing
  Arms: Arm B (informational video); Arm C (informational video and patient navigation)

SUMMARY:
SURGE aims to increase equity in clinical trial enrollment by addressing barriers to genomic testing, which is increasingly needed to assess precision clinical trial eligibility and access standard precision therapies. The study is an interventional pilot meant primarily to assess the feasibility of the intervention. The intervention is comprised of a patient navigator, text message questionnaire, and informational video.

DETAILED DESCRIPTION:
Supporting UnderRepresented populations in Genomics-based cancer trial Enrollment (SURGE) is a multimodal intervention to address medical literacy and unmet social determinants of health (SDoH) needs as barriers to tumor somatic genomic testing consent among historically underrepresented patients (HUP) diagnosed with advanced solid or hematologic malignancies as a prerequisite to precision therapies and/or clinical trial eligibility. Our key hypothesis is that video-based education with or without 1:1 patient navigation will address medical literacy and unmet SDoH barriers, supporting HUP decision-making about genomic tumor consent. We will conduct a type 1 hybrid implementation effectiveness study among a cohort of HUP seeking medical oncology care at two academic and two community practice sites.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 years or older)
* Black, Latinx, OR older adult (age 70 years or older)
* Scheduled for a new patient consultation
* Suspected or confirmed advanced malignancy (requiring active treatment)
* Gastrointestinal, hematologic, or thoracic cancer
* DFCI patient at Longwood/Chestnut Hill, DFCI satellite at St. Elizabeth's Medical Center, or DFCI satellite at Merrimack Valley

Exclusion Criteria:

* Malignancy or former malignancy that requires only surveillance
* Not continuing care at a participating DFCI site
* Speaks a language other than English or Spanish
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Genomic testing uptake | Up to 90 days of enrollment
  Intervention impact on rate of uptake of genomic testing

SECONDARY OUTCOMES:
Patient interaction with the intervention | Up to 30 days of enrollment
  Interaction with each component of the intervention (as appropriate by intervention arm)
Acceptability of questionnaire modality | Up to 30 days of enrollment
  We will use the System Usability Scale to measure usability of the questionnaire electronic tool. The 10-item System Usability Scale is scored on a five-point Likert scale, with 1 being Strongly Disagree and 5 being Strongly Agree.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine J McCleary, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Dana-Farber Cancer Instiute - Merrimack Valley, Methuen, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu